CLINICAL TRIAL: NCT04218097
Title: Impact of Follow-up in Subjects With Obesity and Food Addiction
Brief Title: Food Addiction and Follow-up in Subjects With Obesity
Acronym: ADDICTAL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0401
Record Dates: First submitted 2019-12-19; First posted 2020-01-06 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Eating Disorders; Food Addiction
MeSH Terms: conditions — Obesity; Feeding and Eating Disorders; Food Addiction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Addict patients: Obese type 2 and 3 with food addict according to the Yale Food Addiction Scale (YFAS) questionnaire.
  Cohort design: identification of patients treated in hospital for obesity assessment over the period 1 January 2017 to 1 January 2018 whose addictive or non-addictive status was characterised by the YFAS questionnaire. To talk about food addiction, the person must have at least 3 out of 7 positive criteria AND also meet the "marked suffering" criterion.
  Interventions: Other: Study questionnaire
- Control patients: Obese type 2 and 3, non food addict Cohort design: identification of patients treated in hospital for obesity assessment over the period 1 January 2017 to 1 January 2018 whose addictive or non-addictive status was characterised by the YFAS questionnaire. To talk about food addiction, the person must have at least 3 out of 7 positive criteria AND also meet the "marked suffering" criterion.
  Interventions: Other: Study questionnaire

INTERVENTIONS:
Other: Study questionnaire — Monitoring - data collection: Sending of an information form and the study questionnaire, the YFAS and Hospital Anxiety and Depression (HAD) scale by post within a follow-up period of 24 to 36 months. With a stamped envelope for the answer and a telephone reminder if necessary.

SUMMARY:
Obesity is a chronic disease. Its prevalence, which is constantly increasing, as well as the morbidity and mortality caused, require the development of new treatments, particularly for associated eating disorders. Indeed, it has been shown that a participation of abnormalities of food addiction type behaviour was frequently found in patients hospitalized for obesity (25% of patients). These disorders require specific management if you want to achieve a good weight result. The aim of the study is to compare the weight evolution of patients with addiction-type disorder (addict) versus those without addiction (non-addict) as well as the management modalities.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients grade 2 and 3
* Hospitalized in Endocrinology A from January 1, 2017 to January 1, 2018
* Over 18 years of age
* Not objecting to its participation

Exclusion Criteria:

* No understanding of French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients grade 2 and 3, Hospitalized in Endocrinology A from January 1, 2017 to January 1, 2018
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Weight change: difference between the current weight reported in a questionnaire and the weight measured at the end of hospitalization | month 36
  Evaluate the weight evolution of patients according to their addictive or non-addictive nature, 24-36 months after their discharge from hospital, in Endocrinology for initial obesity assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Martine LAVILLE, PR, Study Director — Hospices Civils de Lyon
Locations (1):
- Service Endocrinologie, Hôpital Lyon Sud,, Pierre-Bénite, France